CLINICAL TRIAL: NCT00960492
Title: A Phase 1 Dose Finding Study of the Safety and Pharmacokinetics of XL184 Administered Orally in Combination With Temozolomide and Radiation Therapy in the First Line Treatment of Subjects With Glioblastoma
Brief Title: Safety Study of XL184 (Cabozantinib) in Combination With Temozolomide and Radiation Therapy in the Initial Treatment of Adults With Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XL184-002
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Glioblastoma; Giant Cell Glioblastoma; Gliosarcoma
Keywords: Astrocytic tumor; Glioblastoma with oligodendroglial components
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Astrocytoma | interventions — Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): XL184 will be initiated at the start of the 6-7 week concurrent phase of RT (+TMZ; some subjects found to have specific gene activity in their tumor tissue may not receive TMZ), given as a single agent during the rest phase (4 weeks), if applicable, and continued subsequently in the maintenance phase.
  Interventions: Drug: XL184; Drug: temozolomide; Radiation: Radiation Therapy
- Arm 2 (Experimental): XL184 will be initiated during the maintenance phase with TMZ
  Interventions: Drug: XL184; Drug: temozolomide
- MTD Expansion (Experimental): XL184 will be initiated at the start of the 6-7 week concurrent phase of RT (+TMZ; some subjects found to have specific gene activity in their tumor tissue may not receive TMZ), given as a single agent in the rest phase (4 weeks), if applicable, and continued subsequently in the maintenance phase. Subjects in this group will receive XL184 and TMZ at the maximally tolerated dose levels determined in Arms 1 and 2.
  Interventions: Drug: XL184; Drug: temozolomide

INTERVENTIONS:
Drug: XL184 — XL184 will be administered daily as a single oral agent supplied as 25- and 100-mg capsules
Drug: temozolomide — TMZ will be supplied as 5-, 20-, 100-, 250-, 140-, and 180-mg capsules. The starting dose will be 75 mg/m2/day given daily with concurrent RT for 6 weeks
  Other Names: Temodar®
  Arms: Arm 1
Drug: temozolomide — TMZ will be supplied as 5-, 20-, 100-, 250-, 140-, and 180-mg capsules. The starting dose will be 200 mg/m2/day given for 5 consecutive days and repeated every 28 days.
  Other Names: Temodar®
  Arms: Arm 2
Radiation: Radiation Therapy — Subjects will receive RT consisting of fractionated focal irradiation administered using 1.8-2 Gy/fraction, daily for 5 days/week for 6-7 weeks, for a total dose of up to 60 Gy.
  Arms: Arm 1
Drug: temozolomide — TMZ will be supplied as 5-, 20-, 100-, 250-, 140-, and 180-mg capsules.
  Other Names: Temodar®
  Arms: MTD Expansion

SUMMARY:
The purpose of this study is to determine the highest safe dose of XL184 administered orally in combination with temozolomide (TMZ, Temodar®) and radiation therapy (RT). XL184 is a new chemical entity that inhibits VEGFR2, MET, and RET, kinases implicated in tumor formation, growth and migration. Temozolomide (TMZ, Temodar®) is an orally administered alkylating agent. It is approved by the Food and Drug Administration (FDA) for the treatment of newly diagnosed glioblastoma (GB) patients when given in combination with radiation therapy (RT) followed by maintenance treatment. First-line treatment for patients with GB consists of a concurrent phase (6-7 weeks in duration) during which TMZ is given with RT, followed by a rest phase (4 weeks in duration; to allow for recovery from delayed toxicity, if present), and a maintenance phase, during which patients receive TMZ for approximately twelve 28-day cycles. To determine the highest safe dose, subjects will receive different amounts of XL184 at different times according to the phase of TMZ and radiation therapy. The first group of subjects will receive the lowest dose of XL184. As long as no medically unacceptable side effects are noted, the dose will be increased for the next group. If the dose is not well-tolerated by the first group of subjects, the dose will be lowered for the next group.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of Grade 4 astrocytic tumor, which includes glioblastoma, giant cell glioblastoma, gliosarcoma, and glioblastoma with oligodendroglial components.
* Must have had a partial or complete surgical resection of the Grade 4 astrocytic tumor.
* Subjects in Arm 1 must have had no previous treatment except surgery (ie, no previous RT, local chemotherapy, or systemic therapy). Subjects must meet certain other eligibility requirements.
* Subjects in Arm 2 must have completed a standard first line regimen of concurrent TMZ and RT for newly diagnosed GB, followed by a rest phase, and has not had any other previous treatment except surgery (including any other regimens of RT and local or systemic chemotherapy). Subjects must meet certain other eligibility requirements.
* Subjects must be able to undergo serial MRIs (computerized tomography [CT] may not substitute for magnetic resonance imaging [MRI]).
* Must be ≥ 18 years old.
* Must have a Karnofsky performance status of ≥ 70% and the ability to swallow whole capsules
* Must have no other diagnosis of malignancy (except surgically excised non-melanoma skin cancer or carcinoma in situ of the cervix, treated early stage prostate cancer, or a malignancy diagnosed ≥ 2 years previously with no current evidence of disease and no therapy within two years prior to enrollment on this study).
* Must be capable of understanding and complying with the protocol requirements and has signed the informed consent document.
* Sexually active fertile subjects (male and female) must agree to use accepted methods of contraception during the course of the study and for 3 months after the last dose of study drug(s).
* Female subjects of childbearing potential must have a negative pregnancy test at screening.

Exclusion Criteria:

* Subject has received prior systemic chemotherapy or RT (Arm 1) or prior systemic chemotherapy other than TMZ (Arm 2), biologic agents, or any other type of investigational agent for the treatment of brain tumors. Subjects who have progressed on TMZ are not eligible.
* Subject has evidence of acute intracranial or intratumoral hemorrhage > Grade 1 either by MRI or CT scan. Subjects with resolving hemorrhage changes, punctate hemorrhage, or hemosiderin may enter the study.
* Subject has serious intercurrent illness such as: hypertension despite optimal treatment, or significant cardiac arrhythmias; or a recent history of serious disease such as symptomatic congestive heart failure, or abdominal fistula or gastrointestinal (GI) perforation within 6 months, prior to starting study treatment.
* Subject has had major surgery within 28 days prior to starting study treatment, or had non water-tight dural closure during previous surgery, or has unhealed wounds from previous surgery.
* Subject has inherited bleeding diathesis or coagulopathy with the risk of bleeding.
* Subject is pregnant or breastfeeding.
* Subject is known to be positive for the human immunodeficiency virus (HIV) (a test for HIV at screening is not required).
* Subject has a previously-identified allergy or hypersensitivity to components of either the XL184 or TMZ formulations.
* Subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-09; Primary Completion 2012-11 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of oral administration of XL184 added to first-line treatment for subjects with newly diagnosed GB | Assessed at every visit to the study clinic
Determine the maximum tolerated dose (MTD) of oral XL184 when added to the concurrent phase of treatment with TMZ and RT and when added to the maintenance phase of treatment with TMZ for subjects with newly diagnosed GB | Assessed periodically as subjects are dose-escalted
Determine the safety and tolerability of XL184 when administered in combination with first-line treatment throughout the concurrent, rest and maintenance phases in an expanded MTD cohort | Assessed at each visit to the study center

SECONDARY OUTCOMES:
Evaluate the plasma pharmacokinetics of XL184 and TMZ when XL184 is administered in combination with TMZ, and of XL184 when it is administered alone, in subjects with newly diagnosed GB | Assessed at 4 visits during the concurrent phase, 2 visits during the first maintenance phase cycle, and approximately every 4 weeks thereafter
Evaluate the pharmacodynamic effects of XL184 (with or without TMZ) and RT in the first line treatment of subjects with GB. | Assessed at 4 visits during the concurrent phase, 2 visits during the first maintenance phase cycle, and approximately every 4 weeks thereafter
Evaluate the preliminary efficacy of XL184 (with or without TMZ) and RT in the MTD expansion cohort in the first line treatment of subjects with GB | Assessed at 10 weeks and approximately every 4 weeks thereafter

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - UCLA, Los Angeles, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Beth Israel Medical Center, New York, New York
  - Duke University Medical Center; The Preston Robert Tisch Brain Tumor Center, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Health System/Division of Neuro-Oncology, Charlottesville, Virginia
  - University of Washington, Seattle, Washington